CLINICAL TRIAL: NCT05909124
Title: A Retrospective Study to Evaluate the Feasibility and Safety of Magnetically Controlled Capsule Endoscope System in Gastric Examination in Obese People
Brief Title: MCE for Gastric Examination in Obese People
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Other Study IDs: MCE for obese people
Record Dates: First submitted 2023-03-30; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy weight people (18.5≤BMI<25): 18.5≤BMI<25
  Interventions: Device: MCE
- obese people (BMI≥30): BMI≥30
  Interventions: Device: MCE

INTERVENTIONS:
Device: MCE — underwent MCE examination

SUMMARY:
This retrospective study aimed to evaluate the feasibility and safety of MCE for the detection of gastric disease in obese people.

DETAILED DESCRIPTION:
In this study, we evaluated the feasibility and safety of MCE for the detection of gastric disease in obese people by comparing the results of MCE between healthy weight people (18.5≤BMI<25) and obese people (BMI≥30). The observation index included mucosal visualization, gastric transit time, cleanliness of the stomach, detection of lesions and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18.5≤BMI<25 or BMI≥30
* underwent gastric examination;
* At least 18 years old；
* Be able to provide informed consent.

Exclusion Criteria:

* With swallowing obstruction or disorders;
* With known or suspected gastrointestinal obstruction, stenosis and fistula;
* Have no conditions for surgery or refuse to undergo any abdominal surgery;
* Be allergic to or have other known contraindication or intolerance to the drug used in the study;
* With pacemakers or other electronic devices such as electronic cochlear implants, implanted magnetic metal drug infusion pumps, neurostimulators, and magnetic metal foreign bodies;
* Women during pregnancy;
* Currently enrolled in another clinical trial of a drug or device;
* Other conditions determined by the investigator to be inappropriate for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18.5≤BMI<25 or BMI≥30；underwent gastric examination; At least 18 years old；Be able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
the degree of gastric mucosal visualization | 2 weeks
  The overall observational integrity of the gastric mucosa is based on the evaluation of the mucosal visualization of several key anatomical sites in the stomach: cardia, fundus, gastric body, gastric horn, gastric antrum and pylorus. The evaluation criteria for mucosal visualization of each site are: good : adequate observation, ≥90% of the gastric mucosa can be observed; fair : good observation, 70-90% of the gastric mucosa can be observed; poor : inadequate observation, <70% of the gastric mucosa can be observed.

SECONDARY OUTCOMES:
the cleanliness of the stomach | 2 weeks
  The criteria for judging the cleanliness of the stomach are: excellent : no adhesive mucus and foam, clear field of view; good : a small amount of mucus and foam, but the field of view is not blurred and does not affect the integrity of the examination; average : medium amount of mucus and foam, the field of view is more blurred and affects the integrity of the examination; poor : a large amount of mucus and foam, the field of view is blurred and affects the integrity of the examination.
Stomach transmit time | 2 weeks
  The time of the first stomach image, the first small intestine image and the last image taken by capsule endoscopy were recorded. Stomach transmit time: time of first small intestine image minus time of first stomach image.
Small bowel transmit time | 2 weeks
  The time of the first large intestine image minus the time of the first small intestine image.
Incidence of adverse events | 2 weeks
  The rates of adverse events such as asphyxia by capsule aspiration, swallow disorder, retention, technical failure, and procedural adverse events were recorded.
Gastric distention | 2 weeks
  Assess condition of gastric distention. The criteria for judging gastric distention is: excellent, no obvious gastric folds; good, moderate distance between gastric folds, without folding; fair, short distance between gastric folds, with small amount of folding; poor, no obvious distance between gastric folds, with large amount of folding

CONTACTS AND LOCATIONS:
Overall Officials: Yangyang Qian, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Liao Z, Duan XD, Xin L, Bo LM, Wang XH, Xiao GH, Hu LH, Zhuang SL, Li ZS. Feasibility and safety of magnetic-controlled capsule endoscopy system in examination of human stomach: a pilot study in healthy volunteers. J Interv Gastroenterol. 2012 Oct-Dec;2(4):155-160. doi: 10.4161/jig.23751. Epub 2012 Oct 1. PMID 23687601
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Background] Zou WB, Hou XH, Xin L, Liu J, Bo LM, Yu GY, Liao Z, Li ZS. Magnetic-controlled capsule endoscopy vs. gastroscopy for gastric diseases: a two-center self-controlled comparative trial. Endoscopy. 2015 Jun;47(6):525-8. doi: 10.1055/s-0034-1391123. Epub 2015 Jan 15. PMID 25590177